# Study Title: Quantifying the Efficacy and Role of Service Dogs for Military Veterans With PTSD

Sponsor: Dr. Marguerite E. O'Haire

ClinicalTrials.gov ID: NCT03245814

Document date: July 20, 2023

# **Brief Summary**

The purpose of this study is to quantify the therapeutic efficacy and role of trained service dogs on socioemotional functioning among military veterans with posttraumatic stress disorder (PTSD).

# **Detailed Description**

The long-term research goal is to evaluate the safety and efficacy of service dogs as a complementary intervention to enhance biopsychosocial functioning in special populations. The objective is to conduct a methodologically rigorous trial to quantify the therapeutic efficacy of service dogs on clinically important outcomes for veterans with PTSD. Based on preliminary findings and qualitative reports, the central hypothesis is that military veterans with PTSD who are provided service dogs will experience reduced PTSD symptoms related to socioemotional functioning and arousal modulation. The rationale for this research is that its successful completion will provide an evidence-based demonstration of the efficacy and role of an increasingly used yet poorly tested complementary intervention. The completion of this project is expected to establish an initial demonstration of the therapeutic efficacy of service dogs in this population, as well as possible mechanisms of action via specific biological pathways and human-canine interaction profiles.

<u>Conditions:</u> Posttraumatic Stress Disorder (PTSD) <u>Intervention / Treatment:</u> Behavioral: Service Dog

#### **Funding**

This work was supported by the Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) and the National Center for Complementary and Integrative Health (NCCIH) of the National Institutes of Health (NIH) under award number R21HD091896, Merrick PetCare and the Dogtopia Foundation. The content is solely the responsibility of the authors and does not necessarily represent the official views of the National Institutes of Health.

# **Participant Criteria**

# Eligibility Criteria

Inclusion criteria for veterans into the study will include:

- Applied for and approved to receive a dog from K9s For Warriors
- Military service on or after September 11, 2001
- Honorable discharge or current honorable service
- Diagnosis of PTSD
- No conviction of any crimes against animals.
- 18 Years and older

# **Study Plan**

Study Design

Primary Purpose: Supportive Care Allocation: Non-Randomized

Interventional Model: Parallel Assignment Masking: Single (Outcomes Assessor)

*Masking Description:* Clinician Administered PTSD Scale for DSM-V (CAPS-5) assessments will be completed via telephone by a trained CAPS-5 rater who will be masked to the intervention and treatment arm of each participant.

# Arms and Interventions

| 11 ms with 1 mc remitals | |
|---|---|
| Participant / Group Arm | Intervention / Treatment |
| Experimental: Service Dog | Behavioral: Service Dog |
| Participants in the service dog arm will receive unrestricted, | A service dog trained to perform tasks that are |
| non-study usual care, in addition to a trained service dog. | specific to PTSD |
| No Intervention: Waitlist Control | |
| Participants in the control arm will receive unrestricted, non- | |
| study usual care, while on the waitlist for a service dog. | |

#### **Outcome Measures**

# **Primary**

| <b>Outcome Measure</b> | Measure Description | Time Frame |
|---|---|---|
| PTSD severity | Posttraumatic Stress Disorder Checklist for DSM-V (PCL-5) | 3 months |
| and symptoms via | | |
| self-report | | |
| PTSD severity | Clinician-Administered PTSD Assessment for the Diagnostic and | 3 months |
| and symptoms via | Statistical Manual of Mental Disorders, Fifth Edition DSM-V (CAPS-5) | |
| clinician rating | | |
| Depression | Patient Reported Outcome Measurement Information System (PROMIS) | 3 months |
| | Adult Short Form (SF) v1.0 - Emotional Distress - Depression 8a | |
| Anxiety | Patient Reported Outcome Measurement Information System (PROMIS) | 3 months |
| | Adult Short Form (SF) v1.0 - Emotional Distress - Anxiety 8a | |

# Secondary

| <b>Outcome Measure</b> | Measure Description | Time Frame |
|---|---|---|
| Social isolation | Patient Reported Outcome Measurement Information System (PROMIS) | 3 months |
| | Adult Short Form (SF) v2.0 - Social Isolation 8a | |
| Companionship | Patient Reported Outcome Measurement Information System (PROMIS) | 3 months |
| | Adult Short Form (SF) v2.0 - Companionship 6a | |
| Ability to | Patient Reported Outcome Measurement Information System (PROMIS) | 3 months |
| participate in | Adult Short Form (SF) v2.0 - Ability to Participate in Social Roles and | |
| social activities | Activities 8a | |
| Mental health | Veterans Rand 12-item Health Survey (VR-12) - Mental Health | 3 months |
| quality of life | Component | |
| Psychological | Bradburn Scale of Psychological Wellbeing (BSPW) | 3 months |
| well-being | | |
| Life satisfaction | Satisfaction with Life Scale (SLS) | 3 months |
| Resilience | Connor-Davidson Resilience Scale (CDRS) | 3 months |
| Anger | Patient Reported Outcome Measurement Information System (PROMIS) | 3 months |
| | Adult Short Form (SF) v1.1 - Emotional Distress - Anger 5a | |
| Daily socio- | Ecological momentary assessment (EMA) | 3 months |
| emotional | - , , , | |
| experiences | | |

# Other Pre-specified

| Outcome Measure | Measure Description | Time Frame |
|---|---|---|
| Work and activity | Work Productivity and Activity Impairment Questionnaire (WPAIQ) | 3 months |
| participation | | |
| Suicidal ideation | Columbia Suicide Severity Rating Scale (CSSRS) | 3 months |
| Sleep quality | Pittsburgh Sleep Quality Assessment (PSQI) | 3 months |
| Sleep disturbance | Patient Reported Outcome Measurement Information System (PROMIS) | 3 months |
| | Adult Short Form (SF) v1.0 - Sleep Disturbance 8a | |
| Sleep actigraphy | Actiwatch 2 (Philips Respironics) | 3 months |
| Salivary cortisol | Passive drool method (Salimetrics) | 3 months |
| awakening | | |
| response | | |
| Electrodermal | Embrace wristband (Empatica, Inc.) | 3 months |
| activity (skin | | |
| conductance) | | |

# **Collaborators and Investigators**

Sponsor: Marguerite O'Haire

#### Collaborators

- Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
- National Center for Complementary and Integrative Health (NCCIH)

# Investigators

• Principal Investigator: Marguerite O'Haire, Ph.D., Purdue University

# Statistical Analysis Plan

Since all the outcome measures are ordinal in nature (based on questionnaire scores), cumulative probability models will be used for all outcomes. While many of these outcomes have been modeled with linear regression in past studies, statisticians have cautioned that treating ordinal data as though they were continuous could potentially lead to misleading results, and that even continuous data can be modeled with cumulative probability models to avoid assumptions about the conditional distribution of the outcome (1,2). Cumulative probability models enable estimation of effect ratios (e.g., veterans allocated service dogs had a lower odds of greater CAPS-5 score compared to veterans on the waiting list), exceedance probabilities (e.g.  $Prob[PHQ-9 \ge 10 \mid X=service dog)$ ), and differences in exceedance probabilities (e.g. absolute risk reduction between veterans allocated a service dog vs control).

In addition to a binary variable for intervention (1=service dog, 0=control), covariates will include the baseline value of the modeled outcome, age, gender/sex, concurrent evidence-based treatment for PTSD, pet ownership, military sexual trauma, and traumatic brain injury.

We will conduct sensitivity analyses, modeling the primary outcomes with ordinary least squares regression to see if our conclusions are sensitive to the model choice, by comparing the estimated conditional means and 95% confidence intervals.

In exploratory analyses, we will consider a potential interaction between treatment and baseline PTSD severity, as baseline severity could modify the effect of service dog.

Multiple imputation will be used for missing covariate data and missing data at the 3-month follow-up visit.

# Software

R package <u>rms</u> (orm function) or <u>rmsb</u> package (blrm function)

# Reporting

- 1. Estimated conditional median (or mean) (e.g., conditional mean PCL-5 given service dog, and given no service dog), with nonparametric bootstrap 95% confidence intervals; adjusted for pre-specified covariates.
- 2. Estimated parameter comparing service dog group to no service dog group (e.g. odds ratio for logit link) with nonparametric bootstrap 95% confidence interval; adjusted for pre-specified covariates.
- 3. For established clinically important cutoffs, exceedance probabilities (Prob[Y ≥ y | X]) will be reported (e.g., Prob[PHQ-9 ≥ 10 | X=service dog]), and differences in exceedance probabilities with nonparametric bootstrap 95% confidence intervals; adjusted for pre-specified covariates.

# References

- 1. <u>Liddell, T. M., & Kruschke, J. K. (2018). Analyzing ordinal data with metric models: What could possibly go wrong?</u>. *Journal of Experimental Social Psychology*, 79, 328-348.
- 2. Liu, Q., Shepherd, B. E., Li, C., & Harrell Jr, F. E. (2017). Modeling continuous response variables using ordinal regression. *Statistics in medicine*, *36*(27), 4316-4335.